CLINICAL TRIAL: NCT05256537
Title: IIT2021-11-PAQUETTE-OmitMMF: Fludarabine and Total Body Irradiation 800 cGy or 1125 cGy For Allogeneic Stem Cell Transplant Using Graft Versus Host Disease Prophylaxis With Post-Transplant Cyclophosphamide and Tacrolimus, Without Mycophenolate Mofetil
Brief Title: Fludarabine and Total Body Irradiation 800 Centigray (cGy) or 1125 cGy For Allogeneic Stem Cell Transplant Using Graft Versus Host Disease Prophylaxis With Post-Transplant Cyclophosphamide and Tacrolimus, Without Mycophenolate Mofetil
Acronym: OmitMMF
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ronald Paquette (Other)
Responsible Party: Sponsor-Investigator, Ronald Paquette, Medical Director, Blood and Marrow Transplant Program, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021-11-PAQUETTE-OmitMMF
Record Dates: First submitted 2022-01-27; First posted 2022-02-25 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Hematologic Neoplasms
Keywords: allogeneic stem cell transplant
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Open-label safety trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Arm (Experimental): Omission of the drug mycophenolate mofetil
  Interventions: Other: Omission of the drug mycophenolate mofetil

INTERVENTIONS:
Other: Omission of the drug mycophenolate mofetil — Elimination of the immunosuppressive drug mycophenolate mofetil (MMF) from the post-transplant regimen.

SUMMARY:
This is a pilot study to evaluate the feasibility, safety and potential benefits of removing one immune suppressive drug called mycophenolate mofetil (MMF) from the standard allogenic stem cell transplant treatment protocol.

MMF will be omitted from the transplant regimen in 60 eligible patients with hematologic malignancies. Participants will be followed for up to 2 years post standard of care transplant at Cedars-Sinai.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18-75 years
* Patient has a related donor who is at least Human Leukocyte Antigen (HLA) haploidentical, or an unrelated donor who is a most a single HLA antigen mismatch.
* Patient signs the Informed Consent Form for the study
* Patient has a hematologic malignancy other than myelofibrosis and meets standard criteria for allogeneic stem cell transplant.
* Patient is deemed suitable to receive Fludarabine and Total Body Irradiation (Flu/TBI) 1125 or Flu/TBI 800 conditioning regimen as standard of care transplant
* Donor is willing to donate peripheral blood stem cells

Exclusion Criteria:

* Patient has a diagnosis of myelofibrosis
* Patient has high titer antibodies against one or more donor HLA antigens
* Patient has undergone prior autologous or allogeneic stem cell transplant.
* Inability to collect sufficient peripheral blood stem cells from the donor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2026-03-07 (Estimated)

PRIMARY OUTCOMES:
Engraftment failure | 60 days post-transplant
  Evaluate the feasibility of eliminating the drug Mycophenolate Mofetil (MMF) from the transplant regimens as determined by an acceptable rate of engraftment failure (<10%). Engraftment failure is when the blood-forming cells received on transplant day do not start to grow and make healthy blood cells.

SECONDARY OUTCOMES:
Time to neutrophil and platelet engraftment | 60 days post-transplant
  Days to neutrophil and platelet engraftment since transplant.
Rate of severe acute GVHD by day +100. | 100 days post-transplant
  Proportion of patients with severe acute GVHD at day 100 post-transplantation.
  * Acute GVHD is when the donated stem cells attack the body within the first 100 days post-transplant.
  * The modified Keystone criteria will be used for acute GVHD staging and grading.
Treatment-related mortality | 5 days post- transplant to 2-years
  Rate of treatment-related mortality
Rate of severe chronic GVHD at 1 year | 1-year post-transplant
  Proportion of patients with severe chronic GVHD at day 365 post-transplantation.
  -Chronic GVHD is when the donated stem cells attack the body after 100 days post-transplant. Chronic GVHD is defined by NIH Consensus Criteria for chronic GVHD.
Relapse | 1 year post-transplant and 2 years post-transplant
  Relapse rate at 1 and 2 years
Overall Survival (OS) | 1-year post-transplant and 2-years post-transplant
  Overall survival at 1 and 2 years
Graft Versus Host Disease (GVHD)-free, Relapse Free Survival | 1-year post- transplant and 2-years post-transplant
  Rate of GVHD-free, Relapse Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Paquette, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States